CLINICAL TRIAL: NCT01619111
Title: DETECT III - A Multicenter, Randomized, Phase III Study to Compare Standard Therapy Alone Versus Standard Therapy Plus Lapatinib in Patients With Initially HER2-negative Metastatic Breast Cancer and HER2-positive Circulating Tumor Cells
Brief Title: DETECT III - A Multicenter, Phase III Study to Compare Standard Therapy +/- Lapatinib in HER2-ve MBC-Patients With HER2+ve CTCs
Acronym: DETECT III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, Prof. Dr. med. Wolfgang Janni, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DETECT III; 2010-024238-46 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-14 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: HER2-negative Metastatic Breast Cancer; HER2-positive Circulating Tumor Cells
Keywords: metastatic breast cancer; circulating tumor cells; lapatinib
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard therapy (Active Comparator): standard chemo- or endocrine therapy
  Interventions: Drug: standard chemo- or endocrine therapy
- standard therapy + lapatinib (Experimental): standard chemo- or endocrine therapy + lapatinib
  Interventions: Drug: standard chemo- or endocrine therapy + Lapatinib

INTERVENTIONS:
Drug: standard chemo- or endocrine therapy — standard chemo- or endocrine therapy:
  * Monochemotherapy (containing one of the following): docetaxel, paclitaxel, vinorelbine, capecitabine, NPLD (non-pegylated liposomal doxorubicin)
  * Endocrine therapy: aromatase inhibitors (anastrozole, letrozole, exemestane)
  Arms: standard therapy
Drug: standard chemo- or endocrine therapy + Lapatinib — Lapatinib
  + standard chemo- or endocrine therapy:
  * Monochemotherapy (containing one of the following): docetaxel, paclitaxel, vinorelbine, capecitabine, NPLD (non-pegylated liposomal doxorubicin)
  * Endocrine therapy: aromatase inhibitors (anastrozole, letrozole, exemestane)
  Arms: standard therapy + lapatinib

SUMMARY:
The HER2 status in breast cancer patients may change during the course of the disease. In 30% of initially HER2-negative patients with circulating tumor cells (CTC), HER2-positive CTCs can be detected in peripheral blood samples(1). At present, it is unclear if therapy based on the HER2 status of CTC offers a clinical benefit for these patients. The DETECT III - trial compares lapatinib, as HER2-targeted therapy in combination with standard therapy versus standard therapy alone in those patients, with initially HER2-negative metastatic breast cancer and HER2-positive circulating tumor cells.

As one of the first interventional trials based on the assessment of CTC phenotypes, the DETECT III - trial aims to evaluate the efficacy of HER2-targeted therapy in patients with MBC and HER2-positive CTCs as well as the significance of CTC as an early predictive marker for treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in study participation.
2. Metastatic breast cancer which cannot be treated by surgery or radiotherapy only. The primary tumor and/or biopsies from metastatic sites or locoregional recurrences must have been confirmed as cancer by histopathology. Estrogen Receptor (EG) and Progesterone Receptor (PgR) status must have been documented.
3. Primary tumor tissue and/or biopsies from metastatic sites or locoregional recurrences were investigated for HER2 status and all of the investigations showed HER2-negativity (i.e.: immunohistochemistry (IHC) score 0-1+ or 2+ and fluorescent in situ hybridization (FISH) negative or just FISH negative, whichever was performed).
4. Evidence of HER2-positive CTCs. Evidence is assumed if the following holds:

   * At least one CTC could be extracted from 7.5 ml patient blood by means of the CellSearch® Circulating Tumor Cell Kit (Veridex LLC) and
   * At least one of all extracted CTCs was found to be HER2-positive. HER2 status must be assessed by means of IHC or FISH.
5. Indication for a standard chemo- or endocrine therapy whose combination with lapatinib is either approved (see SPC of Tyverb® 250 mg tablets) or has been investigated in prior clinical trials (see tables of section 8.2.1.).
6. Tumor evaluation has been performed within 6 weeks before randomization and results are available.
7. Patients must have at least one lesion that can be accurately measured according to RECIST guideline version 1.1 [Eisenhauer 2009].
8. Age ≥ 18 years.
9. ECOG Score < 2
10. Adequate organ function within 7 days before randomization, evidenced by the following laboratory results below:

    * absolute neutrophil count ≥ 1500/µL,
    * platelet count ≥ 100000/µL,
    * hemoglobin ≥ 9 g/dL,
    * ALT (SGPT) ≤ 2.5 × ULN,
    * AST (SGOT) ≤ 2.5 × ULN,
    * serum alkaline phosphatase ≤ 2.5 × ULN, (Serum alkaline phosphatase may be > 2.5 × ULN only if bone metastases are present and AST (SGOT) and ALT (SGPT) < 1.5× ULN)
    * creatinine ≤ 2.0 mg/dl or 177µmol/L
    * International normalized ratio (INR) and activated partial thromboplastin time or partial thromboplastin time (aPTT or PTT) ≤ 1.5 × ULN Please note: These laboratory criteria only refer to lapatinib therapy; with respect to the standard anticancer therapy the relevant summaries of product characteristics (SPCs) have to be observed additionally.
11. Left ventricular cardiac ejection fraction (LVEF) ≥ 50%, in case of planned standard chemotherapy with anthracyclines ≥ 55%, and in any case within normal institutional limits as measured by echocardiogram
12. In case of patients of child bearing potential:

    * Negative pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to randomization,
    * Contraception by means of a reliable method (i.e. non-hormonal contraception, IUD, a double barrier method, vasectomy of the sexual partner, complete sexual abstinence). Patient must consent in maintaining such contraception until 28 days after completion of study treatment.

Exclusion Criteria:

1. History of hypersensitivity reactions attributed to compounds of similar chemical or biological composition to lapatinib.
2. History of > 3 chemotherapy lines for metastatic disease (a chemotherapy line being defined as any new chemotherapy and any modification of an existing chemotherapy regimen regardless of the reason for change).
3. Treatment with investigational agents of any type or anticancer therapy during the trial or within 4 weeks prior to randomization and 6 weeks in case of nitrosoureas or mitomycin C.
4. Adverse events due to prior anticancer therapy which are > Grade 1 (NCI CTCAE) at time of randomization.
5. Anti-retroviral therapy due to HIV infection.
6. Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
7. Concurrent disease or condition that might interfere with adequate assessment or evaluation of study data, or any medical disorder that would make the patient's participation unreasonably hazardous.
8. Other malignant diseases within the last 3 years apart from CIN of the uterine cervix and skin basalioma.
9. Disease or condition which might restrain the ability to take or absorb oral medication. This includes malabsorption syndrome, requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption (for example resection of small bowel or stomach), uncontrolled inflammatory GI disease (e.g., Crohn's disease) and any other diseases significantly affecting gastrointestinal function as well as inability to swallow and retain oral medication for any other reason.
10. Active cardiac disease, defined as:

    * History of uncontrolled or symptomatic angina,
    * history of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation,
    * myocardial infarction less than 6 months from study entry,
    * uncontrolled or symptomatic congestive heart failure,
    * ejection fraction below the institutional normal limit,
    * any other cardiac condition, which in the opinion of the treating physician would make this protocol unreasonably hazardous for the patient.
11. Dementia, altered mental status, or any psychiatric or social condition which would prohibit the understanding or rendering of informed consent or which might interfere with the patient's adherence to the protocol.
12. Life expectancy < 3 months.
13. Male patients.
14. Pregnancy or nursing.
15. Primary tumor or biopsies from metastatic sites or locoregional recurrences showing HER2-positivity.
16. Any prior treatment with anti-HER2 directed therapy.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-02; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
CTC clearance rate | 8 - 12 weeks
  CTC clearance rate: Proportion of patients with at least one CTC detected in 7.5 ml of peripheral blood drawn before treatment that show no evidence of CTCs in the blood after treatment (CTC prevalence as assessed using the Cell-Search® System; Veridex LLC, Raritan, USA)

SECONDARY OUTCOMES:
Overall response rate | 8-12 weeks
  Rate of complete (CR) and partial responses (PR) in patients with whom target lesions were defined
Clinical benefit rate | 8-12 weeks
  Rate of patients who were assessed PR or CR or who had stable disease (SD) for at least 6 months.
Overall survival | 4 weeks
  Time from randomization until death of any cause
Dynamic of CTC | 8-12 weeks
  Descriptive statistics of regular CTC counts
Quality of life (QoL) | 4 weeks
  As assessed by evaluation of the EORTC QLQ-C30 and EORTC QLQ-BR23 questionnaires.
Safety and tolerability of lapatinib | 4 weeks
  Assessed by evaluation of adverse event (AE) reports.
Intensity of pain | 4 weeks
  Measured by use of numeric rating scale (NRS)
Progression free survival (PFS) | 8 - 12 weeks
  Time interval from randomization until progressive disease (PD) or death from any cause, whichever comes first
Level of compliance to study protocol. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Fehm, MD, PhD, Principal Investigator — Heinrich-Heine University, Duesseldorf; Wolfgang Janni, MD, PhD, Study Director — University Hospital Ulm
Locations (1):
- University Hospital Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Fehm T, Muller V, Aktas B, Janni W, Schneeweiss A, Stickeler E, Lattrich C, Lohberg CR, Solomayer E, Rack B, Riethdorf S, Klein C, Schindlbeck C, Brocker K, Kasimir-Bauer S, Wallwiener D, Pantel K. HER2 status of circulating tumor cells in patients with metastatic breast cancer: a prospective, multicenter trial. Breast Cancer Res Treat. 2010 Nov;124(2):403-12. doi: 10.1007/s10549-010-1163-x. Epub 2010 Sep 22. PMID 20859679
- [Derived] Fehm T, Mueller V, Banys-Paluchowski M, Fasching PA, Friedl TWP, Hartkopf A, Huober J, Loehberg C, Rack B, Riethdorf S, Schneeweiss A, Wallwiener D, Meier-Stiegen F, Krawczyk N, Jaeger B, Reinhardt F, Hoffmann O, Mueller L, Wimberger P, Ruckhaeberle E, Blohmer JU, Cieslik JP, Franken A, Niederacher D, Neubauer H, Pantel K, Janni W; DETECT Study Group. Efficacy of Lapatinib in Patients with HER2-Negative Metastatic Breast Cancer and HER2-Positive Circulating Tumor Cells-The DETECT III Clinical Trial. Clin Chem. 2024 Jan 4;70(1):307-318. doi: 10.1093/clinchem/hvad144. PMID 38175595
- See also: Related Info — http://www.detect-studien.de